CLINICAL TRIAL: NCT06350435
Title: Effects of Prefabricated Foot Orthoses With and Without Metatarsal Pads in People With Central Metatarsalgia: A Randomized Controlled Trial
Brief Title: Effects of Prefabricated Foot Orthoses With and Without Metatarsal Pads on Central Metatarsalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Pamela Youde Nethersole Eastern Hospital (Other)
Responsible Party: Principal Investigator, Chan Fung Ting, Student, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CUHK 2023.569
Record Dates: First submitted 2024-04-01; First posted 2024-04-05 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Metatarsalgia
MeSH Terms: conditions — Metatarsalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental)
  Interventions: Device: Prefabricated foot orthoses (PFO) with metatarsal pads
- Control group (Other)
  Interventions: Device: Prefabricated foot orthoses (PFO) without metatarsal pads

INTERVENTIONS:
Device: Prefabricated foot orthoses (PFO) with metatarsal pads — A pair of prefabricated foot orthoses, each with a metatarsal pad to be affixed underneath
  Other Names: Slimflex® Amber Insoles; Podotech® High Density Metatarsal Pad- Wide Raise SD2121, SD2122, SD2123
  Arms: Experimental Group
Device: Prefabricated foot orthoses (PFO) without metatarsal pads — A pair of prefabricated foot orthoses only
  Other Names: Slimflex® Amber Insoles
  Arms: Control group

SUMMARY:
Compare the effects of prefabricated foot orthoses with and without metatarsal pads on pain intensity in the 2nd to 4th metatarsophalangeal joints, foot and ankle functional abilities as well as the occurrence of plantar callosities among patients with central metatarsalgia.

DETAILED DESCRIPTION:
Metatarsalgia is a common condition that affecting about 10% of the general population. Central metatarsalgia involves pathology of the 2nd to 4th metatarsal and their respective metatarsophalangeal joints. This randomized control trial is designed to compare the effects of prefabricated foot orthoses with and without metatarsal pads on pain intensity, foot and ankle functional abilities as well as the occurrence of plantar callosities.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Complain of foot pain on the 2nd to 4th MTPJs during walking in shoes, rating the pain intensity as ≥ 50mm on the Visual Analogue Scale (VAS);
* Able to be ambulant

Exclusion Criteria:

* Peripheral vascular disease (PVD)
* Neurological dysfunctions or neuromuscular disorders
* Active infection, i.e., cellulitis, osteomyelitis, shingles
* Cognitive impairment
* History of lower limb surgery and currently undergoing rehabilitation
* Active ulceration on foot and ankle
* Current utilization of prescribed insoles

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-01-26 (Actual); Primary Completion 2024-04-18 (Actual); Study Completion 2024-04-18 (Actual)

PRIMARY OUTCOMES:
Pain intensity at the 2nd to 4th metatarsophalangeal joints during walking in shoes on Visual Analogue Scale | Baseline, a follow-up at 4-8 weeks from baseline
  VAS consists of a 100mm-long uninterrupted horizontal line, with 2 verbal description at each end. A score of 0mm represents "no pain" while 100 mm represents "the worst imaginable pain".

SECONDARY OUTCOMES:
Foot and Ankle Outcome Score (FAOS) | Baseline, a follow-up at 4-8 weeks from baseline
  FAOS consists of 42 questions, which are categorized into 5 subdomains: symptoms, pain, activities of daily living, sports and quality of life. Each question id rated on a 5-point Likert scale, ranging from 0 to 4 and subsequently transformed into a normalized score between 0 and 100. A score of 100 indicates absence of symptoms, while a score of 0 indicates the presence of severe symptoms.
Size of callosities and corns on the plantar area of the 2nd to 4th metatarsophalangeal joints | Baseline, a follow-up at 4-8 weeks from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Fung Ting Chan, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Pamela Youde Nethersole Eastern Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No